CLINICAL TRIAL: NCT01616680
Title: Phase II Study to Evaluate the Efficacy of Brentuximab Vedotin in Patients With Steroid-Resistant Acute GVHD
Brief Title: Brentuximab Vedotin in Treating Patients With Steroid-Resistant Acute Graft-Versus-Host Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2589.00; NCI-2012-00921 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-06

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (brentuximab vedotin) (Experimental): Patients receive brentuximab vedotin IV over 30 minutes on days 1, 8, and 15.
  Interventions: Drug: brentuximab vedotin; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: brentuximab vedotin — Given IV
  Other Names: Adcetris; anti-CD30 ADC SGN-35; anti-CD30 antibody-drug conjugate SGN-35; antibody-drug conjugate SGN-35; SGN-35
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
The purpose of this research is to test the safety and efficacy of brentuximab vedotin in patients with acute skin graft-versus-host disease (GVHD)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine whether the complete and partial response rate of steroid-resistant skin GVHD exceeds 25% after administration of brentuximab vedotin.

SECONDARY OBJECTIVES:

I. Evaluate the effect of brentuximab vedotin on the clinical manifestations of acute GVHD of the liver and gastrointestinal tract.

II. Determine the incidence and degree of brentuximab vedotin-related toxicity when administered after allogeneic hematopoietic cell transplantation (HCT).

III. Evaluate cluster of differentiation (CD)30 expression in skin biopsies before and after administration of brentuximab vedotin.

IV. Enumerate CD30 expressing lymphocytes in the blood and measure the concentration of soluble CD30 in serum before and after administration of brentuximab vedotin.

V. Determine whether changes in CD30 expression in skin biopsies or blood lymphocytes or the concentration of CD30 in serum before and after administration of brentuximab vedotin are correlated with changes in skin GVHD stage.

VI. Evaluate pharmacokinetics (PK) of brentuximab vedotin in patients after allogeneic HCT.

OUTLINE: This is a dose escalation study.

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on days 1, 8, and 15.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with steroid-resistant stage 2 or 3 acute GVHD of the skin with or without involvement of other organs; patients must have received initial therapy with prednisone or methylprednisolone at a prednisone-equivalent dose of at least 1.0 mg/kg/day alone or combined with other agents, including psoralen and ultraviolet A (PUVA), with:

  * Flare of rash involving at least 25% of the body surface at any time after starting prednisone for GVHD treatment, OR
  * Rash involving more than 50% of the body surface persisting after at least 1 week of initial treatment, OR
  * Rash involving at least 25% of the body surface persisting after at least 2 weeks of initial treatment
* Concomitant use of steroids is permitted; steroid dose should not have been increased within a week prior to enrollment
* Patient, guardian or legally authorized representative is able and willing to provide informed consent
* Willing to use effective contraception; both women of childbearing potential and men who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days after the last dose of study drug

Exclusion Criteria:

* Prior second-line systemic treatment for GVHD
* Absolute neutrophil count (ANC) < 2000/μL
* Administration of growth factor in order to maintain the ANC > 2000/μL
* Platelet count < 30,000/μL, (unsupported)
* Serum total bilirubin concentration > upper limit of normal (ULN)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3X ULN
* Calculated creatinine clearance < 60 ml/min
* Peripheral neuropathy: clinical total neuropathy score (TNS) score > 2
* Any Grade 3 or higher uncontrolled active infection within 1 week before enrollment
* Bullous formation or desquamation related to GVHD (stage 4 skin GVHD)
* Evidence of recurrent/persistent malignancy by cytogenetics, histology or flow cytometry
* GVHD after donor lymphocyte infusion (DLI)
* Clinical manifestations of chronic skin GVHD
* Women who are pregnant or lactating; women of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (beta-hCG) pregnancy test result within 7 days before the first dose of brentuximab vedotin; woman of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy
* Patients with a known hypersensitivity to brentuximab vedotin
* History of Progressive multifocal leukoencephalopathy (PML)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Partial and complete response rates of steroid-resistant acute skin GVHD following administration of brentuximab vedotin | Up to day 28

SECONDARY OUTCOMES:
Complete and partial response rates of gut and liver acute GVHD after administration of brentuximab vedotin | Up to day 28
Incidence and severity of brentuximab vedotin-related toxicity after allogeneic HCT defined graded according to the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE), Version 4 | Assessed up to day 45

CONTACTS AND LOCATIONS:
Overall Officials: Merav Bar, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States